CLINICAL TRIAL: NCT06475859
Title: The Role of Epigenetic Mechanisms in Stress Intolerance in Patients With Chronic Widespread Pain
Acronym: EPISIP
Status: Completed | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Research Foundation Flanders (Other); KU Leuven (Other)
Responsible Party: Principal Investigator, Jo Nijs, Prof. Dr., Vrije Universiteit Brussel
Other Study IDs: EC-2022-118
Record Dates: First submitted 2024-05-16; First posted 2024-06-26 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Chronic Widespread Pain
Keywords: Chronic Widespread Pain; Epigenetics; Autonomic Nervous System; Stress Intolerance
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, Peripheral blood mononuclear cells (PBMC), Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Women with chronic widespread pain: Women who received the diagnosis of fibromyalgia from a doctor.
  Interventions: Other: Montreal Imaging Stress Test; Other: Relaxation breathing
- Healthy women: Healthy women without any chronic diseases or pain in daily life.
  Interventions: Other: Montreal Imaging Stress Test; Other: Relaxation breathing

INTERVENTIONS:
Other: Montreal Imaging Stress Test — A mental stress test that induces stress via a series of arithmetic tasks participants need to solve in a few seconds.
Other: Relaxation breathing — 3 short sessions (4 minutes) of relaxation breathing

SUMMARY:
Patients with chronic widespread pain (CWP) frequently experience stress intolerance - an exacerbation of symptoms in response to stress. Although it severely affects their quality of life, stress intolerance remains a mystery. Hence, unravelling the mechanisms underlying stress intolerance is crucial to understand CWP pathophysiology and to develop novel treatments. Epigenetic mechanisms hold the potential to provide an answer as they have been found to be altered in patients with CWP at baseline, and in response to stress. However, research on epigenetic mechanisms in CWP is very scarce. Hence, this study aims to address this knowledge gap by assessing stress-induced epigenetic changes in patients with CWP and healthy controls aiming to unravel whether epigenetic mechanisms can help explain stress intolerance. The regulatory role of epigenetic mechanisms will be researched in relation to the activity of enzymes affected by the epigenetic mechanisms, neurophysiological measures, and stress-induced symptom changes in patients with CWP.

DETAILED DESCRIPTION:
The objectives of this project will be tackled by a randomized cross-over study including 44 patients with CWP and 44 healthy controls. Participants are expected to come to the hospital twice and fill in questionnaires at several defined timepoints. Two days before their first visit, participants will complete baseline questionnaires at home via REDCap, which will take approximately one hour. Next, participants will be randomised into Group 1 (undergoing the mental stress test at their first visit and then relaxation breathing) or Group 2 (undergoing relaxation breathing at their first visit and then the mental stress test). During each hospital visit, the participants will be assessed before, during and after the intervention. The Pre-test assessment consists of a blood withdrawal, five short questionnaires, examination of pain thresholds, and neurophysiological measurements. The latter will continue during the intervention, which consists of a mental stress test or relaxation breathing. The Post-test assessment consists of a blood withdrawal, one short questionnaire, examination of pain thresholds, and neurophysiological measurements. Then there are again 2 home-based assessments via REDCap 24h and 7 days after the intervention during which the participants will in 1 or 5 short questionnaires, respectively.

ELIGIBILITY:
Inclusion Criteria:

* female
* age between 18 and 70 years old
* body mass index (BMI) below 30
* inactive lifestyle
* for patients only: received the diagnosis of fibromyalgia

Exclusion Criteria:

* other neurological, endocrine, cardiac, or systemic syndromes
* history of cancer or heart failure
* women that are pregnant or within one year after pregnancy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential study participants will be recruited mainly through online advertisements, but also in hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
DNA methylation of catecholamine-degrading enzymes | At baseline (i.e. before the mental stress test or relaxation breathing), and 20 minutes after the mental stress test and relaxation breathing
  DNA methylation status of catechol-O-methyltransferase (COMT), monoamine oxidase (MAO)-A and MAO-B

SECONDARY OUTCOMES:
Genetic variations in catecholamine-degrading enzymes | At baseline
  COMT: rs4818; rs4680 MAO-A: rs6323; MAOA-uVNTR MAO-B: rs1799836 COMT: rs4818; rs4680 MAO-A: rs6323; MAOA-uVNTR MAO-B: rs1799836 COMT: rs4818; rs4680 MAO-A: rs6323; MAOA-uVNTR MAO-B: rs1799836 COMT: rs4818; rs4680; MAO-A: rs6323; MAOA-uVNTR; MAO-B: rs1799836
Catecholamine levels | At baseline (i.e. before the mental stress test or relaxation breathing), and 20 minutes after the mental stress test and relaxation breathing
  Levels of adrenaline, noradrenaline and dopamine in plasma
Heart rate variability | Continuously starting 10 minutes before until 10 minutes after the mental stress test and relaxation breathing
  Heart rate variability measured continuously using the Polar H10
Blood pressure | At baseline (i.e. before the mental stress test or relaxation breathing), during (3 times with 4 minutes in between) and 10 minutes after the mental stress test and relaxation breathing
  Blood pressure, both systolic and diastolic, measured at specified moments using a digital device
Activity of catecholamine-degrading enzymes | At baseline (i.e. before the mental stress test or relaxation breathing), and 20 minutes after the mental stress test and relaxation breathing
  Activity of the enzymes will be defined in plasma or PBMCs
Symptom severity | At baseline (i.e. before the mental stress test or relaxation breathing), and 10 minutes, 24 hours and 7 days after the mental stress test and relaxation breathing
  Symptom severity which is assessed through the Chronic Fatigue Syndrome Symptom List

OTHER OUTCOMES:
Temperature and pressure pain thresholds | At baseline (i.e. before the mental stress test or relaxation breathing), and 20 minutes after the mental stress test and relaxation breathing
  Pain thresholds for warmth and cold measured with the TSA-II, and pressure measured with a digital algometer on the hand and leg. Pain intensity is reported through a numeric rating scale ranging from 0 (no pain) to 10 (worst pain).
Level of stress | At baseline (i.e. before the mental stress test or relaxation breathing), during (3 times with 4 minutes in between) and 10 minutes, 24 hours and 7 days after the mental stress test and relaxation breathing
  Numeric rating scale ranging from 0 (no stress) to 10 (worst stress) indicating the level of stress

CONTACTS AND LOCATIONS:
Overall Officials: Jo Nijs, PhD, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Vrije Universiteit Brussel - UZ Brussel, Brussels, Brussels Capital, Belgium